CLINICAL TRIAL: NCT06164483
Title: Electrophysiological Studies of Auditory Functions and CSF Analyses in Patients With Multiple Sclerosis
Brief Title: Auditory Functions in Patients With Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: University of Catania (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Arianna Di Stadio, Associate Professor fixed time, University of Catania
Other Study IDs: MSSNHL2023
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Hearing Disorders
MeSH Terms: conditions — Multiple Sclerosis; Hearing Disorders | interventions — Audiometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebro-spinal-fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy patients between 20 and 40 years
  Interventions: Diagnostic Test: Auditory test; Other: CSF sampling
- MS group: Patient with Relapsing Remitting MS age between 20 and 40 years
  Interventions: Diagnostic Test: Auditory test; Other: CSF sampling

INTERVENTIONS:
Diagnostic Test: Auditory test — The patients will perform:
  Pure Tone Auditory test + Tympanometry and Stapedial Reflex
  * Speech Perception test
  * In case of tinnitus: tinnitus questionnaire and acuphenometry
  * DPOAEs
  * ABR
Other: CSF sampling — Cerebrospinal Fluid will be collected by lumbar puncture and analyzed

SUMMARY:
The study will analyze the auditory functions of patients with Multiple Sclerosis using auditory tests like pure tone auditory test, speech perception test, Auditory Brain Response (ABR) and Distortion Product Otoacustic Emission (DPOAE). CSF will be collected by lumbar puncture and analyzed looking for inflammatory markers.

The results of DPOAE and CSF will be correlated to identify statistically significant correlation.

DETAILED DESCRIPTION:
Case-Control study

Tools for patients' selection and inclusion in the study

STEP one

* Full medical records detailed for neurological diseases
* Brain and spinal cord MRI performed 12 months (n1) before and most recent one (n2)
* Lumbar puncture
* Blood test
* Questionnaire for screening hearing disorders
* App for screening hearing loss

STEP two

* Pure Tone Auditory test + Tympanometry and Stapedial Reflex
* Speech Perception test
* In case of tinnitus: tinnitus questionnaire and acuphenometry
* DPOAEs
* ABR

STEP three in case of Hearing impairment

- MRI Tractography

ELIGIBILITY:
Inclusion Criteria

* age >18 and <50,
* no history of hearing loss,
* no psychiatric condition
* no familial history of otosclerosis/deafness/genetic hearing loss
* patients with PD and/or MS.

Exclusion Criteria

* Conductive hearing loss
* stroke < 2 years
* cardiovascular disease non under control
* diabetes
* hypotensive disorders
* alcohol abuse
* recreational drug consumption
* epilepsy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy patients and patients with RRMS
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Auditory functions and correlation with CSF findings | 12 months
  The worsening of the hearing thresholds and DPOAE results will be correlated with the presence of inflammatory elements in the CSF

CONTACTS AND LOCATIONS:
Locations (1):
- Arianna Di Stadio, Catania, Sicily, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 24 months for 12 months